CLINICAL TRIAL: NCT07284888
Title: Practices of Prone Positioning Ventilation in Patients With Moderate-to-Severe ARDS in Intensive Care Units: A Registry-Based Observational Study
Acronym: PPV SAFE
Status: Recruiting | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Ling Liu, Professor, Southeast University, China
Other Study IDs: PPV in ARDS
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ARDS patients received PPV
  Interventions: Other: Prone position ventilation

INTERVENTIONS:
Other: Prone position ventilation — Patients underwent prone positioning while receiving invasive mechanical ventilation

SUMMARY:
Acute respiratory distress syndrome (ARDS) is a major cause of mortality in intensive care units. Prone position ventilation (PPV) is an important component of ARDS management and has been shown to reduce mortality in patients with moderate-to-severe ARDS. However, substantial heterogeneity exists in treatment response to PPV. Previous studies suggest that lung morphology-focal versus non-focal patterns based on chest CT-may influence responses to ventilatory strategies, but whether lung morphology modifies the effect of PPV remains unclear. In addition, the benefits and safety of PPV in patients with acute brain injury (ABI) complicated by ARDS are uncertain. Although PPV improves oxygenation, it may impair cerebral venous drainage and increase intracranial pressure, raising concerns about its use in ABI patients. Evidence from randomized trials in this population is limited and excludes patients with more severe hypoxemia or elevated intracranial pressure.

Furthermore, the optimal duration and termination criteria for PPV are not well established. While PPV improves alveolar recruitment and reduces ventilator-induced lung injury, prolonged PPV may lead to excessive sedation exposure and PPV-related complications. Identifying the appropriate timing to discontinue PPV may help balance clinical benefits and potential harms.This study is a prospective, multicenter registry enrolling patients with moderate-to-severe ARDS. The objectives are: (1) To determine whether lung morphology can guide individualized PPV strategies; (2) To evaluate the effectiveness and safety of PPV in patients with ARDS complicated by acute brain injury; (3) To investigate the optimal timing for termination of PPV through target trial emulation methods.In addition to these core objectives, the study will include other exploratory aims.

ELIGIBILITY:
Inclusion Criteria:

1.Age ≥ 18 years 2. Moderate-to-severe ARDS requiring invasive mechanical ventilation, defined as:

1. PaO₂/FiO₂ ≤ 150 mm Hg,
2. PEEP ≥ 5 cm H₂O,
3. ARDS diagnosed according to the 2023 Global Definition.

Exclusion Criteria:

1.Refusal of informed consent by the patient's legally authorized representative

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Moderate-to-severe ARDS
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
60-day mortality | From inclusion to 28 days
  The proportion of patients who are died within 60 days

SECONDARY OUTCOMES:
28-day mortality | From inclusion to 28 days
  The proportion of patients who are died within 28 days
Ventilator-free days at 28 days | From inclusion to 28 days
  Days alive without endotracheal intubation and invasive mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, School of Medicine, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No